CLINICAL TRIAL: NCT00595413
Title: A Randomised, Double-blind, Placebo Controlled, Multi-centre Phase II Study of Atacicept in Anti-TNFα-naïve Patients With Moderate to Severely Active Rheumatoid Arthritis and an Inadequate Response to Methotrexate
Brief Title: Atacicept in Anti-Tumor Necrosis Factor Alpha-naïve Subjects With Rheumatoid Arthritis (AUGUST II)
Acronym: AUGUST II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EMD Serono (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27905; 2007-002536-29
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Results first posted 2016-02-17 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Atacicept; Adalimumab; Humira®
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — TACI receptor-IgG Fc fragment fusion protein; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Atacicept 150 mg with loading dose (Experimental)
  Interventions: Drug: Atacicept: with loading dose
- Atacicept 150 mg without loading dose (Experimental)
  Interventions: Drug: Atacicept
- Adalimumab (Active Comparator)
  Interventions: Biological: Adalimumab
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo matched to atacicept

INTERVENTIONS:
Drug: Placebo matched to atacicept — Placebo matched to atacicept will be administered subcutaneously twice a week for initial 4 weeks, followed by once a week for subsequent 21 weeks.
  Arms: Placebo
Drug: Atacicept: with loading dose — Atacicept will be administered subcutaneously at a dose of 150 milligram (mg) twice a week for initial 4 weeks as loading dose, followed by 150 mg once a week for subsequent 21 weeks.
  Arms: Atacicept 150 mg with loading dose
Drug: Atacicept — Atacicept will be administered subcutaneously at a dose of 150 mg once a week for 25 weeks.
  Arms: Atacicept 150 mg without loading dose
Biological: Adalimumab — Adalimumab (Humira®) will be administered subcutaneously at a dose of 40 mg every other week for 25 weeks.
  Other Names: Humira®
  Arms: Adalimumab

SUMMARY:
The primary objective of this study is to evaluate the efficacy of atacicept compared to placebo in the treatment of signs and symptoms in a subject population with active rheumatoid arthritis (RA), inadequate response to methotrexate (MTX) and no previous exposure to anti-tumor necrosis factor alpha (anti-TNFalpha) therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects greater than or equal to (>=) 18 years of age at the time of informed consent who have RA satisfying American College of Rheumatology (ACR) criteria with a disease history of at least 6 months
* Subjects must have active disease, defined by >=8 swollen joints (out of 66), >=8 tender joints (out of 68) and CRP >=10 milligram per liter (mg/L) and/or erythrocyte sedimentation rate (ESR) >=28 millimeter per hour (mm/hr), despite treatment with MTX at a dose of >=15 milligram per week (mg/week) for greater than (>) 3 months
* Other protocol-defined inclusion criteria could apply

Exclusion Criteria:

* Inflammatory joint disease other than RA
* Previous or concurrent treatment with any approved or investigational biological compound for RA, including but not restricted to any anti-TNFalpha agents, rituximab, abatacept, tocilizumab, interleukin-1 receptor antagonist (IL-1Ra) and belimumab
* Treatment with disease-modifying anti-rheumatic drug (DMARDs) other than MTX
* Participation in any interventional clinical trial within 1 month before study Day 1
* MTX dose >25 mg/week, prednisone dose >10 mg/day (or equivalent), or change in steroid or non-steroidal anti-inflammatory drug (NSAID) dosing regimen within 28 days before study Day 1
* Immunization with live vaccine or immunoglobulin (Ig) treatment within 28 days before study Day 1 or need for such treatment during the study (including follow-up)
* Any history or presence of active or latent tuberculosis, major infection requiring hospitalization or intravenous anti-infectives within 28 days before study Day 1
* Other major concurrent illness or organ dysfunction as specified in the protocol
* Serum IgG below 6 gram per liter (g/L)
* Known hypersensitivity to atacicept or to any of the components of the formulated atacicept
* Other protocol-defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2007-09; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Serono International SA, an affiliate of Merck KGaA Darmstadt, Germany
Locations (2):
- Please Contact US Medical Information, Rockland, Massachusetts, United States
- Please contact the Merck KGaA Communication Center, Darmstadt, Germany

REFERENCES:
- [Derived] van Vollenhoven RF, Kinnman N, Vincent E, Wax S, Bathon J. Atacicept in patients with rheumatoid arthritis and an inadequate response to methotrexate: results of a phase II, randomized, placebo-controlled trial. Arthritis Rheum. 2011 Jul;63(7):1782-92. doi: 10.1002/art.30372. PMID 21452294
- See also: The European League Against Rheumatism (EULAR) — https://b-com.mci-group.com/Abstract/Statistics/AbstractStatisticsViewPage.aspx?AbstractID=15688

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo matched to atacicept was administered subcutaneously twice a week for initial 4 weeks, followed by once a week for subsequent 21 weeks.
- Atacicept 150 mg With Loading Dose: Atacicept was administered subcutaneously at a dose of 150 milligram (mg) twice a week for initial 4 weeks as loading dose, followed by 150 mg once a week for subsequent 21 weeks.
- Atacicept 150 mg Without Loading Dose: Atacicept was administered subcutaneously at a dose of 150 mg once a week for 25 weeks. Participants also received placebo matched to atacicept subcutaneously once a week during initial 4 weeks for blinding purpose (placebo injections alternating with atacicept injections).
- Adalimumab: Adalimumab (Humira®) was administered subcutaneously at a dose of 40 mg every other week for 25 weeks.
Period: Overall Study
Arm/Group | Placebo | Atacicept 150 mg With Loading Dose | Atacicept 150 mg Without Loading Dose | Adalimumab
Started | 76 | 78 | 78 | 79
Completed | 69 | 73 | 70 | 75
Not Completed | 7 | 5 | 8 | 4
Not completed — Adverse Event | 0 | 2 | 1 | 1
Not completed — Lost to Follow-up | 2 | 2 | 1 | 3
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Other | 5 | 1 | 5 | 0

BASELINE CHARACTERISTICS:
Population: Intention-to-treat (ITT) population included all randomized participants who received at least 1 study treatment dose.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Atacicept 150 mg With Loading Dose | Atacicept 150 mg Without Loading Dose | Adalimumab | Total
Number analyzed (Participants) | 76 | 78 | 78 | 79 | 311
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (10.3) | 53.0 (11.3) | 53.3 (13.2) | 53.3 (11.5) | 53.4 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 65 | 66 | 64 | 259
  Male | 12 | 13 | 12 | 15 | 52

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving American College of Rheumatology 20 Response Based on C-reactive Protein (ACR20-CRP) at Week 26
Description: ACR20-CRP response is defined as greater than or equal to (>=) 20 percent (%) improvement from Baseline in both tender joint counts (based on a total of 68 joints) and swollen joint counts (based on a total of 66 joints) together with >=20% improvement from Baseline in at least 3 of the following 5 measures: 1) participant's assessment of pain; 2) participant's global assessment of disease activity; 3) physician's global assessment of disease activity; 4) participant's assessment of physical function; and 5) acute-phase marker (CRP).
Time Frame: Week 26
Population: ITT population included all randomized participants who received at least 1 study treatment dose.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Atacicept 150 mg With Loading Dose | Atacicept 150 mg Without Loading Dose | Adalimumab
Number analyzed (Participants) | 76 | 78 | 78 | 79
percentage of participants | 46.1 | 44.9 | 57.7 | 70.9

2. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50 Response Based on CRP (ACR50-CRP) at Week 26
Description: ACR50-CRP response is defined as >=50% improvement from Baseline in both tender joint counts (based on a total of 68 joints) and swollen joint counts (based on a total of 66 joints) together with >=50% improvement from Baseline in at least 3 of the following 5 measures: 1) participant's assessment of pain; 2) participant's global assessment of disease activity; 3) physician's global assessment of disease activity; 4) participant's assessment of physical function; and 5) acute-phase marker (CRP).
Time Frame: Week 26
Population: ITT population included all randomized participants who received at least 1 study treatment dose.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Atacicept 150 mg With Loading Dose | Atacicept 150 mg Without Loading Dose | Adalimumab
Number analyzed (Participants) | 76 | 78 | 78 | 79
percentage of participants | 14.5 | 29.5 | 33.3 | 38.0

3. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70 Response Based on CRP (ACR70-CRP) at Week 26
Description: ACR70-CRP response is defined as >=70% improvement from Baseline in both tender joint counts (based on a total of 68 joints) and swollen joint counts (based on a total of 66 joints) together with >=70% improvement from Baseline in at least 3 of the following 5 measures: 1) participant's assessment of pain; 2) participant's global assessment of disease activity; 3) physician's global assessment of disease activity; 4) participant's assessment of physical function; and 5) acute-phase marker (CRP).
Time Frame: Week 26
Population: ITT population included all randomized participants who received at least 1 study treatment dose.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Atacicept 150 mg With Loading Dose | Atacicept 150 mg Without Loading Dose | Adalimumab
Number analyzed (Participants) | 76 | 78 | 78 | 79
percentage of participants | 5.3 | 12.8 | 12.8 | 17.7

4. Secondary Outcome: Percentage of Participants With Good or Moderate European League Against Rheumatism (EULAR) Responses at Week 26
Description: The EULAR response criteria evaluate change in DAS28 scores represented as "good response", "moderate response", or "no response" considering both the current DAS28 score and the observed improvement from baseline. Participants were considered to have "good" or "moderate" EULAR response if at the time of assessment, their DAS28 score was less than or equal to (<=) 5.1 and the improvement from baseline in their DAS28 score was greater than (>) 0.6; or if at the time of assessment, their DAS28 score was >5.1 and improvement from baseline in their DAS28 score was >1.2.
Time Frame: Week 26
Population: ITT population included all randomized participants who received at least 1 study treatment dose.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Atacicept 150 mg With Loading Dose | Atacicept 150 mg Without Loading Dose | Adalimumab
Number analyzed (Participants) | 76 | 78 | 78 | 79
percentage of participants | 59.2 | 64.1 | 67.9 | 81.0

5. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event (AE) was defined as any new untoward medical occurrences/worsening of pre-existing medical condition without regard to possibility of causal relationship. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect.
Time Frame: From the first dose of study drug up to 30 days after the last dose of study drug, assessed up to Week 38
Population: ITT population included all randomized participants who received at least 1 study treatment dose.
Measure: Number; unit: participants
Arm/Group | Placebo | Atacicept 150 mg With Loading Dose | Atacicept 150 mg Without Loading Dose | Adalimumab
Number analyzed (Participants) | 76 | 78 | 78 | 79
participants
  TEAEs | 38 | 49 | 49 | 50
  Serious TEAEs | 2 | 4 | 7 | 3

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to 30 days after the last dose of study drug, assessed up to Week 38
Description: An adverse event (AE) is defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to Baseline during a clinical study with an investigational medicinal product (IMP), regardless of causal relationship and even if no IMP has been administered.
Arm/Group | Placebo | Atacicept 150 mg With Loading Dose | Atacicept 150 mg Without Loading Dose | Adalimumab
Serious Adverse Events (participants affected / at risk) | 2/76 | 4/78 | 7/78 | 3/79
Other Adverse Events (participants affected / at risk) | 23/76 | 27/78 | 24/78 | 22/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=76) | Atacicept 150 mg With Loading Dose (N=78) | Atacicept 150 mg Without Loading Dose (N=78) | Adalimumab (N=79)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 2
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Disseminated tuberculosis (Infections and infestations) | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Sudden cardiac death (General disorders) | 0 | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Knee arthroplasty (Surgical and medical procedures) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=76) | Atacicept 150 mg With Loading Dose (N=78) | Atacicept 150 mg Without Loading Dose (N=78) | Adalimumab (N=79)
Bronchitis (Infections and infestations) | 4 | 5 | 6 | 3
Nasopharyngitis (Infections and infestations) | 6 | 2 | 4 | 5
Upper respiratory tract infection (Infections and infestations) | 2 | 4 | 4 | 6
Pharyngitis (Infections and infestations) | 1 | 3 | 4 | 3
Sinusitis (Infections and infestations) | 0 | 5 | 1 | 0
Fatigue (General disorders) | 1 | 2 | 1 | 4
Headache (Nervous system disorders) | 3 | 4 | 4 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 4 | 2
Hypertension (Vascular disorders) | 4 | 3 | 2 | 1
Leukopenia (Blood and lymphatic system disorders) | 4 | 1 | 1 | 3
Urinary tract infection (Infections and infestations) | 3 | 4 | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to publishing results, Institution and Principal Investigator (PI) must first provide Sponsor with a copy of proposed publication for review at least 30 days prior to submission. If Institution and PI do not agree to modification, they shall so notify Sponsor and postpone submission for additional 60 days to allow Sponsor to seek legal remedies or file patent applications. There is a need for coordinated approach to any publication of results from sites for any multi-site study.